CLINICAL TRIAL: NCT07241130
Title: Assessment of End-Tidal CO₂ Levels in the Diagnosis and Management of Patients With Pulmonary Embolism
Brief Title: Using End-Tidal CO₂ to Help Diagnose and Monitor Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bugra Kerget, Associate Professor of Pulmonary Medicine, Ataturk University
Other Study IDs: B.30.2.ATA.0.01.00/427
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Embolism Acute
MeSH Terms: interventions — Thrombolytic Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Group 1: High-Risk Pulmonary Embolism (Thrombolysis): Patients presenting with shock or persistent hypotension and receiving systemic thrombolytic therapy.
  Interventions: Other: thrombolytic therapy
- Group 2: Intermediate-High-Risk Pulmonary Embolism (Thrombolysis): Hemodynamically stable patients with RV dysfunction and elevated biomarkers who required thrombolysis.
  Interventions: Other: thrombolytic therapy
- Group 3: Intermediate-High-Risk Pulmonary Embolism (Non-Thrombolysis): Patients meeting intermediate-high-risk criteria but treated with anticoagulation only.
- Group 4: Healthy Controls: Individuals without cardiopulmonary disease and with normal clinical and laboratory findings.

INTERVENTIONS:
Other: thrombolytic therapy — Participants received standard clinical management according to current pulmonary embolism guidelines. No intervention was assigned by the investigators.
  Groups: Group 1: High-Risk Pulmonary Embolism (Thrombolysis); Group 2: Intermediate-High-Risk Pulmonary Embolism (Thrombolysis)

SUMMARY:
Pulmonary embolism (PE) can reduce blood flow in the lungs and impair gas exchange, leading to lower end-tidal carbon dioxide (EtCO₂) levels. This prospective observational study aims to evaluate whether EtCO₂ can help identify high-risk and intermediate-high-risk patients and monitor early treatment response, especially during thrombolytic therapy. A total of 120 participants were included: high-risk PE, intermediate-high-risk PE patients who received thrombolysis, intermediate-high-risk PE patients treated only with anticoagulation, and healthy controls.

The study measured EtCO₂ along with oxygen saturation, heart rate, respiratory rate, perfusion index, and radiological obstruction scores. By comparing these parameters at diagnosis and during the first 24 hours, the study seeks to determine whether EtCO₂ can serve as a simple, noninvasive marker of disease severity and early hemodynamic improvement in patients with acute PE.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older Diagnosis of acute pulmonary embolism confirmed by CT pulmonary angiography (for PE groups) Classified as high-risk or intermediate-high-risk pulmonary embolism according to ESC/ERS 2019 guidelines Ability to provide informed consent For healthy control group: no history of cardiopulmonary disease, coagulation disorders, or acute medical illness

Exclusion Criteria:

Known chronic respiratory diseases significantly affecting EtCO₂ measurement (e.g., advanced COPD, severe asthma, chronic respiratory failure) Active infection, sepsis, or acute complications of malignancy Prior thrombolytic therapy for pulmonary embolism Anatomical or technical limitations preventing reliable nasal capnography Pregnancy Individuals younger than 18 years Inability or refusal to provide informed consent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study included adult patients diagnosed with acute pulmonary embolism who were classified as high-risk or intermediate-high-risk based on hemodynamic status, right ventricular dysfunction, and cardiac biomarker elevation. Participants were consecutively enrolled at a tertiary university medical center. The study also included a healthy control group composed of adults without cardiopulmonary disease or significant medical comorbidities. A total of 120 individuals were studied across four cohorts representing different clinical risk categories and routine treatment pathways.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
End-Tidal Carbon Dioxide (EtCO₂) Level at Diagnosis | At baseline (within first 1 hour of diagnosis)
  EtCO₂ level measured in mmHg using nasal capnography at the time of diagnosis to assess its ability to identify high-risk and intermediate-high-risk pulmonary embolism and to predict the need for thrombolytic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)